CLINICAL TRIAL: NCT02961179
Title: Nutrigenomics Approach to Investigate the Benefits of Dairy Product Consumption on Glucose Homeostasis
Brief Title: Dairy Products, Diabetes and Genetics
Acronym: PRODIGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2017-3228
Record Dates: First submitted 2016-11-03; First posted 2016-11-10 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2018-01

CONDITIONS: Insulin Sensitivity; Type2 Diabetes
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Increased dairy product (Experimental): Subjects will be asked to consume a total of 3 to 5 servings per day.They will be instructed on options and variations for incorporating the dairy foods into their routine dietary pattern.
  Interventions: Behavioral: Increased dairy product
- Dietary counselling (Placebo Comparator): Subjects will review the standard dietary recommendation(http://www.diabetes.ca/diabetes-and-you/nutrition/meal-planning-guide/) by a registered dietitian.
  Interventions: Behavioral: Dietary counselling

INTERVENTIONS:
Behavioral: Increased dairy product
  Arms: Increased dairy product
Behavioral: Dietary counselling
  Arms: Dietary counselling

SUMMARY:
This study will investigate the in-depth the benefits of dairy consumption on glucose metabolism in patients at risk of type 2 diabetes using novel genomics methodology.To do so, 33 individuals at risk of type 2 diabetes will be randomly subjected to an intervention study including a 6-week intensive dairy product consumption period and a 6-week dietary counselling period.

DETAILED DESCRIPTION:
More than 9 million Canadians are living with diabetes or prediabetes. Type 2 diabetes is a disorder characterized by high blood glucose. Dietary modification is a key component in type 2 diabetes management. For example, dairy product consumption has beneficial effects on metabolic health. Yet, researchers have shown that mixed results exists for insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men and postmenopausal women (absence of menstrual cycles for >12 months) aged >18 yrs;
* BMI between 25-40 kg/m2;
* Hyperinsulinemia (fasting plasma insulin >90 pmol/l);
* Fasting plasma glucose (FPG) <7.0 mmol/l; HbA1c <6.5%);
* If treated with lipid-lowering agents, the dose must have been stable over the last 3 months;
* Stable body weight (±5%) for 3 months;
* Willing to consume study foods and able to follow protocol and give informed consent.

Exclusion Criteria:

* Failure to meet any one or more of the inclusion criteria;
* Diagnosis of type 2 diabetes;
* High dairy consumption ( 2 servings/day or more);
* Major surgery in the 3 months prior to study onset;
* Smoking;
* Incompatibility with dairy consumption (allergy, intolerance or dislike);
* Inflammatory bowel disease or other gastrointestinal disorder influencing gastrointestinal motility or nutrient absorption;
* Medications known to affect lipid and glucose metabolism other than those used to treat hypertension or dyslipidemia;
* Diseases known to affect glucose metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 6 weeks in insulin sensitivity between high dairy and dietary counselling phases | Change from 0 to 6 weeks
  2h-oral glucose tolerance test (OGTT)

SECONDARY OUTCOMES:
Change from baseline to 6 weeks in fasting glucose between high dairy and dietary counselling phases | Change from 0 to 6 weeks
Change from baseline to 6 weeks in 2 h plasma glucose post OGTT between high dairy and dietary counselling phases | Change from 0 to 6 weeks
Change from baseline to 6 weeks in insulin secretion (Insulinogenic index ) between high dairy and dietary counselling phases | Change from 0 to 6 weeks
  Insulinogenic index
Change from baseline to 6 weeks in insulin secretion (area under the curve of C-peptide) between high dairy and dietary counselling phases | Change from 0 to 6 weeks
  Area under the curve of C-peptide
Change from baseline to 6 weeks in b-cell function (disposition index) between high dairy and dietary counselling phases | Change from 0 to 6 weeks
Change from baseline to 6 weeks in glucagon-like peptide-1 secretion between high dairy and dietary counselling phases | Change from 0 to 6 weeks
Change from baseline to 6 weeks in fat mass between high dairy and dietary counselling phases | Change from 0 to 6 weeks
  Dual-energy X-ray absorptiometry
Change from baseline to 6 weeks in blood pressure between high dairy and dietary counselling phases | Change from 0 to 6 weeks
Change from baseline to 6 weeks in aortic stiffness (pulse wave velocity) between high dairy and dietary counselling phases | Change from 0 to 6 weeks
Change from baseline to 6 weeks in lipid profile (total-cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides) between high dairy and dietary counselling phases | Change from 0 to 6 weeks
Change from baseline to 6 weeks in inflammatory profile (C-reactive protein, Tumor necrosis factor-alpha, Interleukin-6) between high dairy and dietary counselling phases | Change from 0 to 6 weeks
Change from baseline to 6 weeks in oxidative stress profile (F2-isoprostane profiles) between high dairy and dietary counselling phases | Change from 0 to 6 weeks
Change from baseline to 6 weeks in fatty acid profile between high dairy and dietary counselling phases | Change from 0 to 6 weeks
Change from baseline to 6 weeks in serum 25(OH) vitamin D between high dairy and dietary counselling phases | Change from 0 to 6 weeks
Change from baseline to 6 weeks in gene expression profiles between high dairy and dietary counselling phases | Change from 0 to 6 weeks
Change from baseline to 6 weeks in metabolomics profiles between high dairy and dietary counselling phases | Change from 0 to 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Research Center CHU de Quebec-Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arghavani H, Bilodeau JF, Rudkowska I. Impact of dairy intake on circulating fatty acids and associations with blood pressure: A randomized crossover trial. Nutr Metab Cardiovasc Dis. 2025 Sep;35(9):104112. doi: 10.1016/j.numecd.2025.104112. Epub 2025 Apr 30. PMID 40436701
- [Derived] Khorraminezhad L, Rudkowska I. Modulation of gene expression profile following consumption of high-dairy products in subjects with hyperinsulinemia. Nutr Metab Cardiovasc Dis. 2023 Jan;33(1):219-226. doi: 10.1016/j.numecd.2022.10.015. Epub 2022 Nov 1. PMID 36411217
- [Derived] Khorraminezhad L, Rudkowska I. Dairy Product Intake Modifies MicroRNA Expression among Individuals with Hyperinsulinemia: A Post-Intervention Cross-Sectional Study. Lifestyle Genom. 2022;15(3):77-86. doi: 10.1159/000523809. Epub 2022 Feb 25. PMID 35220313
- [Derived] O'Connor S, Julien P, Weisnagel SJ, Gagnon C, Rudkowska I. Impact of a High Intake of Dairy Product on Insulin Sensitivity in Hyperinsulinemic Adults: A Crossover Randomized Controlled Trial. Curr Dev Nutr. 2019 Jul 24;3(8):nzz083. doi: 10.1093/cdn/nzz083. eCollection 2019 Aug. PMID 31453424